CLINICAL TRIAL: NCT02353247
Title: Use of Norethindrone Acetate for Management of Bleeding Associated With the Etonogestrel Contraceptive Implant
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norton Healthcare (Other)
Responsible Party: Principal Investigator, Scott LaJoie, Principal Investigator, Norton Healthcare
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-N0278
Record Dates: First submitted 2014-12-02; First posted 2015-02-02 (Estimated); Results first posted 2022-03-16 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-02

CONDITIONS: Etonogestrel Contraceptive Implant, Bothersome Bleeding
MeSH Terms: interventions — Norethindrone Acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Norethindrone acetate (aygestin) (Other): Norethindrone acetate (aygestin) will be used to manage bothersome bleeding. Patients will be prescribed aygestin 5 mg by mouth twice daily for one month, followed by aygestin 5 mg by mouth once daily for two months. Medication will then be discontinued. Patients will be evaluated in the office three months after medication initiation, and then again six months after medication initiation. If the patient is unable to take norethindrone acetate (aygestin) due to medical contraindications or cost, they will receive medroxyprogesterone acetate (provera) 10 mg once daily as alternate oral progesterone. Figure 1 below highlights the study
  Interventions: Drug: Norethindrone acetate

INTERVENTIONS:
Drug: Norethindrone acetate
  Other Names: Aygestin

SUMMARY:
The overall objective of this study is to confirm that oral progesterone is an effective way to manage bothersome bleeding; thus increasing the rate of continuation of the etonogestrel contraceptive implant in adolescents.

DETAILED DESCRIPTION:
The investigators will conduct a prospective study of adolescents using the etonogestrel contraceptive implant. Participants will be recruited from the Kosair Children's Hospital Gynecology Specialists practice in Louisville, Kentucky. This practice provides care to a diverse population of females, from a wide range of socioeconomic statuses, age birth to 25 years.

All patient presenting and choosing to have an implant placed will be offered participation. All enrollments will be voluntary. Participants will not receive compensation for their participation. After obtaining informed consent and assent, participants will provide baseline demographic information, including: age, race/ethnicity, zip code of residence, health insurance provider, number of current and past partners, use of prior contraceptive methods, concomitant condom use, sexually transmitted infection history,smoking status, weight and height. The date of etonogestrel implant insertion will be confirmed.

All patients using etonogestrel contraceptive implants will receive daily SMS texts in the evening via the Qualtrics SMS program asking them to respond with their bleeding pattern that day. The investigators will record responses according to the World Health Organization definitions of bleeding: (a) bleeding day, (b) spotting day, (c) bleeding--- free day [see Table I for WHO bleeding definitions]. At their initial follow---up visit 3 months after Nexplanon insertion, the investigators will identify those who report "bothersome" bleeding patterns. For the purpose of this study, "bothersome" bleeding will be defined as prolonged and/or frequent bleeding, as characterized by World Health Organization---recommended definitions of bleeding. The definitions are listed in Table I.

Bleeding day Any day with vaginal discharge containing blood that required more than 1 sanitary pad or tampon per day

Spotting day Any day with vaginal discharge containing blood that required at most one sanitary pad or tampon per day Bleeding---free day A day during which neither bleeding nor spotting was reported

Bleeding--- spotting episode One or more consecutive days during which bleeding or spotting was entered in the diary, bounded by bleeding---free days

Amenorrhea No bleeding or spotting days throughout the 90---day reference period

Infrequent bleeding Less than three bleeding---spotting episodes in a 90---day reference period, excluding amenorrhea

Normal frequency Three to five bleeding---spotting episodes in a 90---day reference period

Frequent bleeding More than five bleeding---spotting episodes in a 90---day reference period

Prolonged bleeding Any bleeding---spotting episode (uninterrupted) lasting more than 14 days in the 90---day reference period

Table I: WHO bleeding descriptions and patterns

Norethindrone acetate (aygestin) will be used to manage bothersome bleeding. Patients will be prescribed aygestin 5 mg by mouth twice daily for one month, followed by aygestin 5 mg by mouth once daily for two months. Medication will then be discontinued. Patients will be evaluated in the office three months after medication initiation, and then again six months after medication initiation. If the patient is unable to take norethindrone acetate (aygestin) due to medical contraindications or cost, they will receive medroxyprogesterone acetate (provera) 10 mg once daily as alternate oral progesterone. Figure 1 below highlights the study design.

Contraceptive implant inserted & enrollment in the study

Bleeding patterns recorded via SMS text x 3 months

Office visit

Normal bleeding pattern Bothersome bleeding pattern

Continue to record bleeding pattern Aygestin 5 mg PO BID x 1 month*

Continue to record bleeding pattern Aygestin 5 mg PO daily x 2 months

Continue to record bleeding pattern No mediation x 3 months

Office visit Office visit

*Or provera 10 mg PO daily x 3 months

Figure 1: Study design

During the aygestin administration, patients will again receive daily SMS texts in the evening via the Qualtrics SMS program asking them to respond with their bleeding pattern that day. The investigators will record responses according to the World Health Organization definitions of bleeding: (a) bleeding day, (b) spotting day, (c) bleeding--- free day. Patients not reporting bothersome bleeding after the initial 90 days will continue to record bleeding via SMS texts for the next 6 months to serve as the control group (normal bleeding group).

All completed demographic data collection forms and electronic menstrual calendars will be kept in a database, de---identified, and stored on a password--- protected computer. Study size will be a convenience sample. Based on the current rate of etonogestrel implant insertions in our practice, it is anticipated that 30 participants can be recruited over a six---month period of time.

Data Collection and Analysis

All patients who meet the inclusion criteria and enroll in the study will be sent a text message daily for 90 days (3 months). The daily message will prompt the participant to indicate the bleeding level for the day. This single question will have 4 options:

1. Bleeding Day
2. Spotting Day
3. Bleeding Free Day
4. Prefer not to answer today.

On day 90, descriptive tallies of the responses will be done. Using SPSS v20, an algorithm will count the number of bleeding days, spotting days, and bleeding free days and prefer not to answer (PNA) days; the data record for each participant will contain four count variables (bleeding, spotting, free, PNA). Secondly, the algorithm will identify and tally -according to WHO guidelines in Table 1 --- bleeding---spotting episodes (BSE),amenorrhea (AM), infrequent bleeding (IF), normal frequency of bleeding (NF), frequent bleeding (FB), and prolonged bleeding (PB).

Participants who have at least a single episode of FB or PB will be assigned the label of "bothersome bleeding". Those without a single episode of FB or PB will be labeled "normal bleeding". Participants in the Bothersome Bleeding group will be offered aygestin to control the bothersome bleeding. Participants in the Normal Bleeding group will continue as before, with no additional medications. Following the principle of intent---to---treat, data from those in the Bothersome Bleeding group will be assigned to the aygestin group, despite that they are not taking it. During the first month, participants in the Bothersome Bleeding group will take one 5 mg tablets of aygestin twice daily (morning and evening). After 30 days, the dose of aygestin will be halved, such that only one 5 mg tablet is taken daily. Sixty days later, the Bothersome Bleeding group will discontinue aygestin. Ninety days later, both the normal group and the Bothersome Bleeding group will be re-evaluated.

Data Analysis

A descriptive table will be used to sort participants into Normal Bleeding and Bothersome Bleeding. Non---parametric and parametric statistics will be used to compare the demographics of these two groups.

A dose---response curve covering six months will be plotted for the Bothersome Bleeding group to visually reveal the impact of one month of 10 mg of aygestin vs. two months of 5 mg aygestin vs. three months 0 mg of aygestin. Plotted on the curve will be the group averages of the daily bleeding value (1 for no bleeding, .5 for spotting, 0 for bleeding). A second no---dose curve will be added to the X---Y plot for the six months of data from the Normal Bleeding group.

Repeated Measure Multivariate Analysis of Variance (RM---ANOVA) with a Between--- Subjects variable included, will be conducted (assuming sufficient data is available - e.g., low PNA rates) to compare the first 30 day average bleeding value, the 90 day bleeding average, and the 180 day bleeding average between the two groups. Planned post---hoc comparisons will evaluate changes between the control group and intervention group at the three time points. Additional analyses may also include regression analysis to assess for predictive factors related to response to aygestin.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria will include any post---menarchal female presenting to the Kosair Children's Hospital Gynecologic Specialist practice, who desires to use the etonogestrel contraceptive implant and has access to a mobile phone device.

Exclusion Criteria:

* NA

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2017-06-29 (Actual); Study Completion 2017-06-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott LaJoie, PhD, Principal Investigator — University of Louisville
Locations (1):
- Kosair Children's Hospital, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Study Arm: Intervention Group
- Control Group: No intervention
- Consented, Never Randomized: For various reasons (e.g., lost phone access), never responded to initial text survey. As a result, they were not randomized to groups nor tracked during study. Baseline data was collected immediately after consenting.
Period: Overall Study
Arm/Group | Study Arm | Control Group | Consented, Never Randomized
Started | 30 | 23 | 35
Completed | 21 | 18 | 0
Not Completed | 9 | 5 | 35

BASELINE CHARACTERISTICS:
Groups:
- No Intervention (Completed); Intervention (Complete): Completed the full study (at least 70%)
- No Intervention (Did Not Complete): Took med off protocol Responded to less than 70% of text messages
- Intervention (Did Not Complete): Non compliant with medication Requested medication off protocol
- Consented, Never Assigned to Group: Reasons include:
  Minimal response, no show to visit Never responded, no show to visit Technical difficulties Desired to be off all medications Loss of phone privileges Never Got Texts Cell# Changed Too Busy Unknown
- Total: Total of all reporting groups
Arm/Group | No Intervention (Completed) | No Intervention (Did Not Complete) | Intervention (Complete) | Intervention (Did Not Complete) | Consented, Never Assigned to Group | Total
Number analyzed (Participants) | 18 | 5 | 21 | 9 | 35 | 88
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.78 (2.13) | 17.33 (.57) | 15.24 (1.55) | 16.17 (.98) | 16.25 (2.02) | 15.93 (1.88)
Sex: Female, Male [Count of Participants; unit: Participants] — Note, this study only enrolled females.
  Participants
    Female | 18 | 5 | 21 | 9 | 35 | 88
    Male | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 5 | 5 | 5 | 15 | 33
  White | 15 | 0 | 16 | 4 | 18 | 53
  More than one race | 0 | 0 | 0 | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 1
BMI [Mean (Standard Deviation); unit: kg/m^2] | 25.63 (6.32) | 27.19 (8.26) | 26.97 (7.18) | 27.62 (5.57) | 26.41 (5.81) | 26.50 (6.22)
Insurance [Count of Participants; unit: Participants]
  Private | 7 | 2 | 7 | 1 | 12 | 29
  Public | 11 | 2 | 12 | 5 | 23 | 53
  Unknown | 0 | 1 | 2 | 3 | 0 | 6
# Lifetime Sexual Partners [Mean (Standard Deviation); unit: Partners] | .93 (1.1) | 3.33 (4.04) | .59 (.62) | 3.83 (4.62) | 1.69 (1.53) | 1.52 (2.03)
Age of Menarche [Mean (Standard Deviation); unit: years] | 12 (1.14) | 12 (1.00) | 11.52 (1.21) | 12.67 (1.21) | 11.25 (1.92) | 11.61 (1.57)

OUTCOME MEASURES:

1. Primary Outcome: Impact of Aygestin (and Dose of Aygestin) on the Management of Bothersome Bleeding Associated With the Etonogestrel Contraceptive Implant
Description: "Bothersome bleeding" was defined per WHO classification as either frequent bleeding (greater than 5 bleeding-spotting episodes in a 90-day reference period) or prolonged bleeding (any bleeding-spotting episode, uninterrupted, lasting greater than 14 days in a 90-day reference period)
  The scale used was derived from the WHO classification system:
  Bleeding Day (assigned value = 1) Spotting Day (assigned value = .5) Bleeding Free Day (assigned value = 0) Prefer not to answer today (assigned value = missing)
  Higher scores (average of the time period) indicate more bothersome bleeding; low scores indicate less bothersome bleeding. Less bothersome bleeding is the desired outcome.
  Note, the scale is not a published scale but rather was constructed for this study.
Time Frame: Initial 3 months of baseline collection (medicine free); For intervention group, 3 months of medicine, followed by 3 months of medicine free; For control group, 6 months of medicine free.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Control Group T1: Medicine free (months 1-3)
- Control Group T2: Medicine free (months 4-6)
- Control Group T3: Medicine free (months 7-9)
- Intervention Group T1: Reported bothersome bleeding, medicine free (months 1-3)
- Intervention Group T2: Reported bothersome bleeding, prescribed acetate (months 4-6)
- Intervention Group T3: Reported bothersome bleeding, medicine free (months 7-9)
Arm/Group | Control Group T1 | Control Group T2 | Control Group T3 | Intervention Group T1 | Intervention Group T2 | Intervention Group T3
Number analyzed (Participants) | 18 | 18 | 18 | 21 | 21 | 21
units on a scale | 2.73 (.20) | 2.77 (.26) | 2.76 (.24) | 2.27 (.33) | 2.65 (.33) | 2.67 (.27)

ADVERSE EVENTS:
Time Frame: 9 months *data collected every three months
Groups:
- Control Group T1: Did not receive medication (months 1-3)
- Control Group T2: Did not receive medication (months 4-6)
- Control Group T3: Did not receive medication (months 7-9)
- Intervention Group T1: Reported bothersome bleeding, prescribed acetate (months 1-3)
- Intervention Group T3: Reported bothersome bleeding, prescribed acetate (months 7-9)
Arm/Group | Control Group T1 | Control Group T2 | Control Group T3 | Intervention Group T1 | Intervention Group T2 | Intervention Group T3
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/18 | 0/18 | 0/21 | 0/21 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18 | 0/18 | 0/21 | 0/21 | 0/21
Other Adverse Events (participants affected / at risk) | 0/18 | 0/18 | 0/18 | 0/21 | 0/21 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-11-14): https://cdn.clinicaltrials.gov/large-docs/47/NCT02353247/Prot_000.pdf
  • Statistical Analysis Plan (2016-11-14): https://cdn.clinicaltrials.gov/large-docs/47/NCT02353247/SAP_001.pdf